CLINICAL TRIAL: NCT07270406
Title: Healthy Behaviors for Insomnia Prevention in People With HIV and Ongoing Pain
Acronym: HIP HOP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Burel Goodin, Professor of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202508064; R01MD021001 (NIH)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Insomnia; HIV
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Behavioral Treatment for Insomnia (BBTI) (Experimental): BBTI is comprised of four, 30-min weekly sessions, each of which will be administered via telephone. BBTI, utilizes two critical behavioral principles: sleep restriction and stimulus control.
  Interventions: Behavioral: Brief Behavioral Treatment for Insomnia (BBTI)
- Brief Mindfulness Training (BMT) (Experimental): Brief Mindfulness Training (BMT) is comprised of four, 30-min weekly sessions, each of which will be delivered via telephone. BMT utilizes concepts of being aware of what the body is sensing and feeling in the moment in order to achieve a state of calmness and relaxation.
  Interventions: Behavioral: Brief Mindfulness Training (BMT)

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment for Insomnia (BBTI) — BBTI is comprised of four, 30-min weekly sessions, each of which will be administered via telephone. BBTI, utilizes two critical behavioral principles: sleep restriction and stimulus control.
  Arms: Brief Behavioral Treatment for Insomnia (BBTI)
Behavioral: Brief Mindfulness Training (BMT) — Brief Mindfulness Training (BMT) is comprised of four, 30-min weekly sessions, each of which will be delivered via telephone. BMT utilizes concepts of being aware of what the body is sensing and feeling in the moment in order to achieve a state of calmness and relaxation.
  Arms: Brief Mindfulness Training (BMT)

SUMMARY:
The purpose of this research study is to test whether Brief Behavioral Treatment for Insomnia (BBTI) delivered over the phone or Brief Mindfulness Training (BMT) delivered over the phone is better able to improve the symptoms of insomnia, reduce chronic pain, and slow the pace of biological aging in individuals with HIV and Chronic Pain.

ELIGIBILITY:
Inclusion Criteria

Each subject must meet all of the following criteria and be confirmed with electronic medical records:

1. Confirmed HIV diagnosis and currently a patient in the WashU Infectious Disease Clinic
2. Age 25-65 years
3. All people with HIV must be currently receiving stable antiretroviral therapy
4. People with HIV with insomnia must report Insomnia Severity Index >/= 15 at initial screening and meet DSM-5 diagnostic criteria for insomnia including sleep difficulty that occurs at least 3 times per week and has been a problem for at least 3 consecutive months
5. People with HIV must also report the presence of chronic pain on the Brief Chronic Pain Screening Questionnaire and rate their chronic pain as >/= 3 on a 0-10 scale of intensity.

Exclusion Criteria

Subjects will not be enrolled if any of the following criteria exist and confirmed with electronic medical records:

1. History of stroke in past 12 months
2. Active cancer with treatment
3. Heart disease
4. Uncontrolled hypertension
5. Epilepsy
6. Active pregnancy
7. Reynaud's disease
8. Traumatic injury or surgical procedure within the last 12 months
9. Acute infection as suggested by thermometry temperature >100.4
10. Serious psychiatric disorder (bipolar disorder, psychotic disorder)
11. Active suicidal ideation
12. Evidence for severe obstructive sleep apnea (AHI >30/hr) according to Home Sleep Monitoring or presence of another sleep disorder other than insomnia (i.e., not insomnia) as indicated by SCISD-R

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-01-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
sleep quality as determined by the Insomnia Severity Index (ISI) | 4 months
  Sleep quality as determined by the Insomnia Severity Index (ISI), a brief screening tool for insomnia, seven-item questionnaire that asks respondents to rate the nature and symptoms of their sleep problems using a Likert-type scale.
  Scoring:
  Add the scores for all seven items (questions 1 + 2 + 3 + 4 + 5 +6 + 7) = _______ your total score
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
pain severity and interference (BPI-SF). | 4 months
  Pain severity and interference as measured by the Brief Pain Inventory - Short Form, (BPI-SF), a self-administered questionnaire designed to assess both the severity of pain and its impact on daily function.
  Scoring:
  Pain Severity Score = Mean of items 3-6 (pain at its worst, pain at its least, average. Higher scores indicate greater pain severity, range 0-10) Pain Interference Score = Mean of items 9A-9G (interference of pain with: general activity, mood, walking, normal work, relations, sleep, enjoyment of life. Higher scores indicate greater pain interference, range 0-10)

SECONDARY OUTCOMES:
Quality of life (SF-36) | 4 months
  Quality of life as measured by the Short Form - 36, (SF-36), a multi-purpose survey designed to capture adult patients' perceptions of their own health and well-being.
  Scoring: The SF-36 has several scaled scores; the scores are weighted sums of the questions in each section.
  Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability
  The sections of the questionnaire will be broken into two groups, Physical and Mental. The physical section will ask about general health, limitations of activities, pain, and physical health problems. The mental section will ask about emotional health problems, social activities, and energy and emotions.
pace of biological aging (DunedinPACE). | 4 months
  DunedinPACE will allow for a measurement of the rate of biological decline.

CONTACTS AND LOCATIONS:
Overall Officials: Burel Goodin, PhD, Principal Investigator — WashU Medicine

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start date: 12 months following primary outcomes publication End date: No end date
Access Criteria: Any qualified investigator will be able to access all de-identified data upon request and approval by Principal Investigator (Goodin)